CLINICAL TRIAL: NCT01679704
Title: Determination of Glycemic Index (GI) of Ten Food Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Asia Pacific Holdings Pte, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: GIS.2012
Record Dates: First submitted 2012-08-30; First posted 2012-09-06 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-08

CONDITIONS: Glycemic Index
MeSH Terms: interventions — Food

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Food products (Other): Ten food products will be given to all subjects
  Interventions: Dietary Supplement: Food products

INTERVENTIONS:
Dietary Supplement: Food products

SUMMARY:
This study is initiated to investigate the glycemic index value of ten food products.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-pregnant females (at least 6 weeks postpartum, non-lactating)
* Age between 21 to 60 years

Exclusion Criteria:

* Suffering from any chronic diseases.
* Suffering from gastrointestinal diseases that may interfere with nutrient absorption, distribution, metabolism and excretion.
* History of diabtes mellitus or use of antihyperglycemic drugs or insulin to treat diabetes and related conditions.
* History of AIDS, hepatitis, renal or heart disease or any other serious complications that may interfere with glucose metabolism.
* Current use of medication that may interfere with the digestion and nutrient absorption (for examples steriods, protease inhibitors or antipsychotics medications).
* Current use of medication known to affect glucose tolerance (excluding oral contraceptives).
* Known food allergy or intolerance.

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2012-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Glycemic index values of all ten products | 120 minutes post adminstration
  Glycemic index values at 120 minutes post adminstration.

CONTACTS AND LOCATIONS:
Overall Officials: Kalpana Bhaskaran, Dr, Principal Investigator — Temasek Polytechnic
Locations (1):
- Temasek Polytechnic, Singapore, Singapore